CLINICAL TRIAL: NCT07139379
Title: Virtual Reality Multisensory Cooperative Task-Oriented Mirror Therapy for Neuro-Rehabilitation
Brief Title: Effects of Virtual Reality Multisensory Cooperative Task-Oriented Mirror Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-113-307
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Rehabilitation; Virtual Reality; Mirror Movement Therapy; Task Performance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Mirror Therapy Group (Active Comparator): 30 minutes of task-based Virtual Reality Mirror Therapy combined with 20 minutes of conventional task-oriented therapy.
  Interventions: Other: task-oriented training; Other: Virtual Reality Mirror Therapy
- Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Mirror Therapy Group (Experimental): 30 minutes of Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Mirror Therapy combined with 20 minutes of conventional task-oriented therapy.
  Interventions: Other: task-oriented training; Other: Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Mirror Therapy

INTERVENTIONS:
Other: task-oriented training — Motor training targeted to goals that are relevant to the functional needs of the patient
Other: Virtual Reality Mirror Therapy — Virtual Reality Mirror Therapy using goggle
  Arms: Virtual Reality Mirror Therapy Group
Other: Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Mirror Therapy — Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Mirror Therapy using goggle
  Arms: Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Mirror Therapy Group

SUMMARY:
In the proposed study, the investigators assumed that Virtual Reality-Based Generative Bimanual Cooperative Task-Oriented Therapy (VRMCTOMT) will provide a better treatment effects than traditional virtual reality mirror therapy (VRMT) for the patients with unilateral stroke. The aim of the study is to examine the difference in the treatment effects among the combination of task-oriented training with either VRMCTOMT, or VRMT on the upper extremity function and brain activity of the stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke with unilateral side involved;
* A score of Mini-mental state examination greater than 24 for proving higher mental function
* Time of onset > 6 months before treatment begins; and
* Premorbid right-handedness.

Exclusion Criteria:

* Severe vision impairment;
* Major cognitive-perceptual deficit;
* Other brain disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the result of Fugl-Meyer assessment (FMA) for motor function of upper extremity test | baseline, 9 weeks and 21 weeks
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.

SECONDARY OUTCOMES:
Change in the result of Modified Ashworth scale (MAS) | baseline, 9 weeks and 21 weeks
  Muscle tone is defined by the resistance of a muscle being stretched without resistance.

OTHER OUTCOMES:
Change in the result of Box and blocks test | baseline, 9 weeks and 21 weeks
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, 9 weeks and 21 weeks
  The Semmes-Weinstein monofilamenttest examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome.
Change in the result of Motor Activity Log | baseline, 9 weeks and 21 weeks
  Semi-structured interview examine how much and how well the subject uses their more-affected arm for 30 ADLs. Score range from 0-5. Higher values represent a better outcome.
functional Magnetic Resonance Imaging | baseline, 9 weeks
  a non-invasive neuroimaging technique that measures brain activity by detecting changes in blood oxygenation (BOLD signal).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan